CLINICAL TRIAL: NCT02073305
Title: Prognostic Impact of Sleep Apnea on Cardiovascular Morbidity and Mortality, in End Stage Renal Disease Patients
Acronym: SASinHD_003
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Adam Ogna, Centre d'Investigation et Recherche sur le Sommeil (CIRS), Centre Hospitalier Universitaire Vaudois
Other Study IDs: CIRS-SASinHD_003
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea; End Stage Renal Disease
Keywords: obstructive sleep apnea; end stage renal disease; cardiovascular events
MeSH Terms: conditions — Sleep Apnea, Obstructive; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No sleep apnea: Subjects with no or light sleep apnea (AHI < 15/h)
  Interventions: Other: No Sleep Apnea
- Sleep Apnea - untreated: Subjects with moderate to severe sleep apnea (AHI ≥15/h) and no specific treatment.
  Decision to treat or not sleep apnea is left to the treating physician, independently of the study protocol.
  Interventions: Other: Sleep Apnea - untreated
- Sleep Apnea - treated: Subjects with treated moderate to severe sleep apnea (AHI ≥15/h). Decision to treat or not sleep apnea is left to the treating physician, independently of the study protocol.
  Interventions: Device: Sleep Apnea - treated

INTERVENTIONS:
Other: No Sleep Apnea — No intervention
  Groups: No sleep apnea
Other: Sleep Apnea - untreated — No intervention
  Groups: Sleep Apnea - untreated
Device: Sleep Apnea - treated — Sleep Apnea treatment by positive pression ventilation (CPAP/BIPAP) or sleep apnea oral appliance
  Groups: Sleep Apnea - treated

SUMMARY:
The purpose of this study is to prospectively evaluate the impact of sleep apnea on the cardiovascular morbidity and mortality of patients with end-stage renal disease.

DETAILED DESCRIPTION:
Sleep apnea is more prevalent in end stage renal disease patients than in the general population, and may participate to the increased cardiovascular mortality observed in this group of patients. Despite a significant increase in knowledge about the harmful effects of obstructive sleep apnea in the general population, the prognostic impact of sleep apnea in the end stage renal disease population has not yet been investigated.

The purpose of this trial is to investigate the hypothesis that moderate to severe sleep apnea increase the risk of major cardiovascular events in patients with end stage renal disease.

The severity of sleep apnea is measured at inclusion and the patients are followed during 3 years to assess the cardiovascular end-points. The result of the sleep study is communicated to the treating physician and the decision whether to treat or not sleep apnea is left to the treating physician, independently of the study protocol. The comparison will include three groups: patients without sleep apnea, untreated patients with moderate to severe sleep apnea and treated patients with sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease on renal replacement therapy
* age ≥ 18 years

Exclusion Criteria:

* unstable congestive heart failure
* active psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with end stage renal disease on renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Time to first major cardiovascular event | 3 years
  composite end-point of all-cause mortality, acute myocardial infarction, hospitalization for acute myocardial ischemia, acute heart failure, stroke, acute peripheral vascular event

SECONDARY OUTCOMES:
Time to cardiovascular death | 3 years
Time to first non-fatal acute myocardial infarction | 3 years
Time to first hospitalization for acute myocardial ischemia | 3 years
Time to first acute heart failure | 3 years
Time to first non-fatal stroke | 3 years
Time to first acute peripheral vascular event | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Heinzer, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV); Adam Ogna, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV); Valentina Forni Ogna, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland